CLINICAL TRIAL: NCT06245928
Title: Development of an Individualized Respiratory Exercise Device Originated in Turkey and Investigation of Its Clinical Effects on Healthy Individuals
Brief Title: The Effects of Individualized Respiratory Exercise Device in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: buhucgun04
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Respiratory Exercise Device; Biomedical Device; Pulmonary Function; Respiratory Muscle Strength; Functional Capacity; Respiratory Muscle Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The individuals in the experimental group will be trained with an individualized respiratory exercise device for 5 days a week for 8 weeks. The initial pressure load will be set to the resistance level corresponding to 40% of the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements. Participants will be asked to rest following 6 breathing cycles and repeat a total of 36 breathing cycles (6 sets) in each session. Participants will be able to practice both inspiratory and expiratory respiratory muscle training in one breathing cycle. Progression will be increased by 5-10% weekly, with the perceived exertion level being in the range of 4-6 according to the Modified Borg Scale. In addition, physical activity will be recommended.
  Interventions: Device: Individualized Respiratory Exercise Device
- Control Group (Active Comparator): The individuals in the control group will be trained with Threshold® IMT + Threshold™ PEP training for 5 days a week for 8 weeks. Respiratory muscle training will be performed with Threshold® IMT and Threshold™ PEP devices. The training intensity will be set to 40% of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) measurements in the first week. Participants will be asked to perform 6 sets of 6 repetitions for inspiratory and expiratory muscle training separately for a total of 36 repetitions each. Progression will be increased by 5-10% weekly so that the perceived exertion level will be in the range of 4-6 according to the Modified Borg Scale. If the training threshold exceeds the upper-pressure limits of the Threshold® IMT + Threshold™ PEP devices, the training intensity will be continued at the highest limit. In addition, physical activity will be recommended.
  Interventions: Device: Threshold® IMT + Threshold™ PEP

INTERVENTIONS:
Device: Individualized Respiratory Exercise Device — The Individualized Respiratory Exercise device will include both inspiratory muscle training, expiratory muscle training, and intensive spirometer features.
  Arms: Experimental Group
Device: Threshold® IMT + Threshold™ PEP — The Threshold® IMT device allows inspiratory muscle training and the Threshold™ PEP device allows expiratory muscle training.
  Arms: Control Group

SUMMARY:
Respiratory exercise devices can be grouped as respiratory muscle training (RMT) devices and incentive spirometers (IS). IS can improve pulmonary ventilation using visual feedback but cannot increase respiratory muscle strength. RMT devices strengthen the respiratory muscles by their resistance mechanisms but they cannot provide visual feedback. It has been stated that RMT increases exercise performance in healthy individuals. RMT devices usually allow only one of inspiratory muscle training or expiratory muscle training. The need to acquire 2 devices for combined training increases the cost. It is seen that the RMT devices available in Turkey do not allow combined training and a significant part of them do not offer sufficient loading range.

The aims of the project are; to develop a multifunctional individualized respiratory exercise device originating in Turkey, and to analyze the clinical effects of an individualized respiratory exercise device on pulmonary function, respiratory muscle strength, and functional capacity in healthy individuals. The device to be developed in this project will be the first multifunctional respiratory exercise device originated in Turkey. The device will have the clinical features of IS and RMT devices and can be individualized according to the desired purpose. With the same device, the individual will be able to both improve the ventilation of the lungs like the IS and strengthen the respiratory muscles in the direction of inspiration and/or expiration with wide loading intervals.

A total of 46 healthy individuals will be included in the study. The healthy individuals included in the study will be randomly divided into two groups experimental group (n=23) and control group (n=23). The individuals in the experimental group will be trained with an individualized respiratory exercise device for 5 days a week for 8 weeks. The individuals in the control group will be trained with Threshold® IMT + Threshold™ PEP training for 5 days a week for 8 weeks. In both groups, pulmonary function, respiratory muscle strength, and functional capacity will be assessed before and after the 8 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Answering "No" to the general health questions of the Exercise Readiness Questionnaire for all

Exclusion Criteria:

* Being an amateur or professional athlete who does sports-specific training at least 2 times a week
* Having a chronic disease
* Having history of spontaneous or trauma-related pneumothorax
* Having pathologies related to the middle ear (such as tympanic membrane rupture, otitis)
* Receiving routine medical treatment other than vitamin supplements for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | 8 weeks
  Maximal Inspiratory Pressure will be measured in accordance with ATS/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Maximal Expiratory Pressure (MEP) | 8 weeks
  Maximal Expiratory Pressure will be measured in accordance with ATS/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Forced Vital Capacity (FVC) | 8 weeks
  Forced Vital Capacity will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Volume in 1 second (FEV1) | 8 weeks
  Forced Expiratory Volume in 1 second will be measured before six-minute walk test according to the guideline of ERS.
Peak Expiratory Flow (PEF) | 8 weeks
  Peak Expiratory Flow will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Flow 25-75% (FEF25-75) | 8 weeks
  Forced Expiratory Flow 25-75% will be measured before six-minute walk test according to the guideline of ERS.
Spiropalm 6-minute Walk Test | 8 weeks
  The 6-minute Walk Test will be performed with Spiropalm 6 DYT (Cosmed, Spiropalm 6MWT) according to ATS guidelines. Walking distance, minute ventilation, respiratory rate, inspiratory capacity and breathing reserve will be recorded.

SECONDARY OUTCOMES:
Convenience of Device Use | 8 weeks
  A 5-point Likert scale will be used to question the convenience of use of the devices used. Scoring will be determined as 1- "very difficult to use", 5- "very easy to use".

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No